CLINICAL TRIAL: NCT05482243
Title: Protein Supplementation and Exercise Training to Increase Muscle Protein Synthesis Rates in Patients With Advanced Chronic Kidney Disease
Brief Title: Protein and Exercise Training in Chronic KIDNEY Disease
Acronym: PET KIDNEY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: METC 22-032
Record Dates: First submitted 2022-07-28; First posted 2022-08-01 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Kidney Diseases; Muscle Loss
MeSH Terms: conditions — Kidney Diseases; Muscular Atrophy | interventions — Whey Proteins; Resistance Training

STUDY DESIGN:
Intervention Model Description: Randomized crossover study (1-week intervention vs. 1-week habitual lifestyle) for both patients with advanced CKD and healthy controls
Who Masked: Outcomes Assessor
Masking Description: Participants will be randomized to either start with the habitual lifestyle period or the exercise training period. All randomization procedures will be executed by an independent researcher. Due to the nature of the intervention, blinding of participants and investigators during the exercise training period is not possible. During the analysis, the research technicians will only receive the participant codes to ensure blinding during analysis of blood, saliva, and muscle 2H-enrichment. Thereafter, an independent researcher will provided a blinded dataset to the research team.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Habitual lifestyle period (No Intervention): * All participants will be encouraged to keep their diet and physical activity similar to before the study period. Subjects will be asked to record their food intake and wear an Actical physical activity monitor for 3 days throughout the habitual lifestyle period (2 week days and 1 weekend day).
  * All participants will be asked to ingest 20 mL deuterated water and take a saliva sample daily
- Exercise training period (Experimental): * All participants will be encouraged to keep their diet and physical activity similar to before the study period. Subjects will be asked to record their food intake and wear an Actical physical activity monitor for 3 days throughout the exercise training period (2 week days and 1 weekend day).
  * Participants will be asked to ingest 20 mL deuterated water and take a saliva sample daily
  * Participants will visit the University three times with 2-day intervals (e.g. Monday-Wednesday-Friday) for an exercise training session as described in 5.6.
  * Following the training sessions, participants will be provided with a protein supplement as described in 5.7.
  * Before and after ingestion of the protein supplement, participants will be asked to fill in a gastrointestinal tolerance and palatability survey.
  Interventions: Dietary Supplement: Whey protein

INTERVENTIONS:
Dietary Supplement: Whey protein — Throughout 1 week (either in week 1 or 2), all participants will perform a 1-week resistance type exercise-training program, consisting of two different exercises. Leg press and leg extension exercise will be performed on regular weightlifting machines (Technogym, Rotterdam) at 3 days during the 1-week period (e.g. Monday-Wednesday-Friday). During the resistance exercise training protocol, participants will continue their habitual diet as usual. However, patients with CKD will be provided with a protein supplement following the exercise sessions.
  Other Names: Resistance exercise
  Arms: Exercise training period

SUMMARY:
When patients progress to the final stage of chronic kidney disease (CKD) and require hemodialysis treatment, they typically have lost so much muscle function that they are no longer physically independent. However, due to disease- and hemodialysis-related muscle catabolism, dietary protein and exercise interventions are only capable to attenuate the decline in physical function of patients on hemodialysis treatment. Therefore, lifestyle interventions to increase muscle function should be implemented before hemodialysis is required. However, it is still a matter of debate whether muscle protein synthesis rates of patients with advanced CKD can be increased with a patient-tailored dietary protein and exercise intervention.Therefore, the current study will assess MPS rates during habitual lifestyle and during an interventional program including dietary protein and exercise in patients with advanced CKD. In addition, we will compare MPS rates during free-living conditions between patients with advanced CKD and healthy controls.

ELIGIBILITY:
1. In order to be eligible to participate in this study, a patient with CKD must meet all of the following criteria:

   * (e)glomerular filtration rate (GFR) <45 ml/min/1.73m2
   * Age: 18 - 80 y
   * Able to provide written informed consent
2. In order to be eligible to participate in this study, a healthy subject must meet all of the following criteria:

   * (e)GFR >60 ml/min/1.73m2 without albuminuria
   * Age: 18 - 80 y
   * Able to provide written informed consent

1. A potential subject with CKD who meets any of the following criteria will be excluded from participation in this study:

* Insulin-dependent diabetes mellitus or two or more oral glucose lowering medications
* Active inflammatory disease / malignancies
* Uncontrolled hypertension (>160/100mm Hg), unstable angina pectoris, or arrhythmia
* Pulmonary disease restricting exercise performance (e.g. COPD)
* A history of neuromuscular problems
* Cognitive Impairment
* Diagnosed GI tract diseases / dysphagia
* Allergies to milk proteins / Lactose intolerance
* Pregnancy
* Hospitalization <1 months prior to study period
* Participation in any structured exercise program
* Any medications known to affect protein metabolism (i.e. corticosteroids or prescription strength acne medications).
* Use of DOAC, vitamin-K-antagonist, or multiple anticoagulants.
* Dialysis treatment or previous kidney transplantation

  2. A potential healthy subject who meets any of the following criteria will be excluded from participation in this study:
* Insulin-dependent diabetes mellitus or two or more oral glucose lowering medications
* Active inflammatory disease / malignancies
* Uncontrolled hypertension (>160/100mm Hg), unstable angina pectoris, or arrhythmia
* Pulmonary disease restricting exercise performance (e.g. COPD)
* A history of neuromuscular problems
* Cognitive Impairment
* Diagnosed GI tract diseases / dysphagia
* Allergies to milk proteins / Lactose intolerance
* Pregnancy
* Hospitalization <1 months prior to study period
* Participation in any structured exercise program
* Any medications known to affect protein metabolism (i.e. corticosteroids or prescription strength acne medications).
* Use of DOAC, vitamin-K-antagonist, or multiple anticoagulants.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-12-02 (Actual); Study Completion 2024-12-02 (Actual)

PRIMARY OUTCOMES:
Muscle protein synthesis rates | 1-week period
  Muscle protein synthesis rates as measured by the deuterated water method

SECONDARY OUTCOMES:
Physical activity levels | 1-week period
  as measured by accelerometry
Dietary intake (energy/macronutrient) | 1-week period
  as measured by dietary diaries
Leg fat free mass | Baseline
  as measured by DEXA
Body composition | Baseline
  as measured by BIA
Type I and II skeletal muscle fiber size | Baseline
  of muscle biopsy of vastus lateralis
Skeletal muscle mitochondrial bioenergetics | Baseline
  of muscle biopsy of vastus lateralis
Muscle strength | Baseline
  1-RM max testing of leg press and leg extension
Aerobic capacity | Baseline
  VO2-peak test on ergometer

CONTACTS AND LOCATIONS:
Overall Officials: Luc JC van Loon, Prof. Dr., Principal Investigator — Maastricht University
Locations (1):
- Maastricht University Medical Center+, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
Not yet determined